CLINICAL TRIAL: NCT01601470
Title: An Open Label, Three-period, Single Sequence Study to Evaluate the Pharmacokinetic Drug-drug Interaction Between LCZ696 and Sildenafil in Subjects With Mild to Moderate Hypertension
Brief Title: Evaluation of Drug-drug Interaction Between LCZ696 and Sildenafil in Subjects With Mild to Moderate Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CLCZ696B2225; 2012-001632-64 (EudraCT Number)
Record Dates: First submitted 2012-05-16; First posted 2012-05-18 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Mild to Moderate Hypertension
Keywords: LCZ696, sildenafil, pharmacokinetics, mild to moderate hypertension
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Period 1:Sildenafil;Period 2:LCZ696;Period 3:LCZ696+Sildenafil (Experimental): During Treatment Period 1, on study Day 1, participants received a single dose of sildenafil followed by wash out on Day 2. In Period 2 (study Days 3-7), participants received LCZ696 once daily. In Period 3, on study Day 8, participants received LCZ696 , co-administered at the same time with a single dose of sildenafil.
  Interventions: Drug: LCZ696; Drug: Sildenafil

INTERVENTIONS:
Drug: LCZ696 — LCZ696 400mg QD was administered alone for 4 days and in combination with sildenafil for 1 day
Drug: Sildenafil — Sildenafil 50 mg single dose was administered alone for 1 days and in combination with LCZ696 400mg QD for 1 day

SUMMARY:
This study was conducted to investigate the potential for a pharmacokinetic drug-drug interaction in support of the co-administration of LCZ696 and sildenafil.

DETAILED DESCRIPTION:
This study was conducted to investigate the potential for a pharmacokinetic drug-drug interaction in patients with mild-to-moderate hypertension in support of the co-administration of LCZ696 and sildenafil.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with mild to moderate hypertension, either treated or not currently on treatment, between age 18 and 65 years of age, and otherwise in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* At screening: systolic blood pressure 120-140 mmHg on therapy, or 140-160 mmHg if untreated
* At screening: diastolic blood pressure, 70-95 mmHg on therapy, or 90-100 mmHg if untreated
* Baseline: BP ≥140/90;

Exclusion Criteria:

* Use of non-antihypertensive prescription drugs, herbal supplements, and/or over-the-counter (OTC) medication, dietary supplements (vitamins included) within two (2) weeks prior to initial dosing

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Berlin, Germany

REFERENCES:
- [Derived] Hsiao HL, Langenickel TH, Petruck J, Kode K, Ayalasomayajula S, Schuehly U, Greeley M, Pal P, Zhou W, Prescott MF, Sunkara G, Rajman I. Evaluation of Pharmacokinetic and Pharmacodynamic Drug-Drug Interaction of Sacubitril/Valsartan (LCZ696) and Sildenafil in Patients With Mild-to-Moderate Hypertension. Clin Pharmacol Ther. 2018 Mar;103(3):468-476. doi: 10.1002/cpt.759. Epub 2017 Nov 3. PMID 28599060

RESULTS

PARTICIPANT FLOW:
Groups:
- Period 1:Sildenafil;Period 2:LCZ696;Period 3:LCZ696+Sildenafil: During Treatment Period 1, on study Day 1, participants received a single dose of sildenafil followed by a wash out on Day 2. In Period 2 (study Days 3-7), participants received LCZ696 once daily. In Period 3, on study Day 8, participants received LCZ696, co-administered at the same time with a single dose of sildenafil.
Period: Period 1 - Sildenafil
Arm/Group | Period 1:Sildenafil;Period 2:LCZ696;Period 3:LCZ696+Sildenafil
Started | 28
PK Analysis Set | 28
Safety Set | 28
Completed | 28
Not Completed | 0
Period: Period 2 - LCZ696
Arm/Group | Period 1:Sildenafil;Period 2:LCZ696;Period 3:LCZ696+Sildenafil
Started | 28
PK Analysis Set | 27
Safety Set | 27
Completed | 27
Not Completed | 1
Not completed — Physician Decision | 1
Period: Period 3 - LCZ696+Sildenafil
Arm/Group | Period 1:Sildenafil;Period 2:LCZ696;Period 3:LCZ696+Sildenafil
Started | 27
PK Analysis Set | 27
Safety Set | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Period 1:Sildenafil;Period 2:LCZ696;Period 3:LCZ696+Sildenafil
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval (AUCtau) of LCZ696 Analytes
Description: The effect of co-administration of sildenafil on the pharmacokinetics of LCZ696 (analytes of LCZ696: AHU377, LBQ657 and valsartan) was assessed. Blood samples were collected at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose from day 1 to day 7, 24 hours post-dose from day 7, and day 8 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose. AUC is a mathematically-derived value from all measurements. AUC is a measure of the area under the curve that is obtained from plotting the plasma concentration by time point. All time-points were used to derive the single PK parameters.
Time Frame: From pre-dose on day 1 until 12 hours post dose on day 8
Population: PK Analysis Set (Period 3): This set included participants with evaluable PK data and without any protocol deviations which could impact the PK data.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Period 1:Sildenafil;Period 2:LCZ696;Period 3:LCZ696+Sildenafil
Number analyzed (Participants) | 27
h*ng/mL
  AHU377 | 3700 (912)
  LBQ657 | 147000 (31000)
  valsartan | 23600 (9500)

2. Primary Outcome: Maximum Plasma Concentration Following Drug Administration at Steady State (Cmax,ss) of LCZ696 Analytes (AHU377, LBQ657 and Valsartan)
Description: The effect of co-administration of sildenafil on the pharmacokinetics of LCZ696 (analytes of LCZ696: AHU377, LBQ657 and valsartan) was assessed. Blood samples were collected at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose from day 1 to day 7, 24 hours post-dose from day 7, and day 8 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose. Cmax is a mathematically-derived value from all measurements. Cmax is a measure of the area under the curve that is obtained from plotting the plasma concentration by time point. All time-points were used to derive the single PK parameters.
Time Frame: From pre-dose on day 1 until 12 hours post dose on day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Period 1:Sildenafil;Period 2:LCZ696;Period 3:LCZ696+Sildenafil
Number analyzed (Participants) | 27
ng/mL
  AHU377 | 2310 (1020)
  LBQ696 | 14000 (2420)
  valsartan | 3350 (1480)

3. Primary Outcome: Minimum Plasma Concentration Following Drug Administration at Steady State (Cmin,ss) of LCZ696 Analytes (AHU377, LBQ696 and Valsartan)
Description: The effect of co-administration of sildenafil on the pharmacokinetics of LCZ696 (analytes of LCZ696: AHU377, LBQ657 and valsartan) was assessed. Blood samples were collected at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose from day 1 to day 7, 24 hours post-dose from day 7, day 8 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose. Cmin is a mathematically-derived value from all measurements. Cmin is a measure of the area under the curve that is obtained from plotting the plasma concentration by time point. All time-points were used to derive the single PK parameters.
Time Frame: From pre-dose on day 1 until 12 hours post dose on day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Period 1:Sildenafil;Period 2:LCZ696;Period 3:LCZ696+Sildenafil
Number analyzed (Participants) | 27
ng/mL
  AHU377 | 0.0 (0.0)
  LBQ657 | 2170 (733)
  valsartan | 197 (96.9)

4. Primary Outcome: Time to Reach the Maximum Concentration After Drug Administration (Tmax) of LCZ696 Analytes (AHU377, LBQ657 and Valsartan)
Description: The effect of co-administration of sildenafil on the pharmacokinetics of LCZ696 (analytes of LCZ696: AHU377, LBQ657 and valsartan) was assessed. Blood samples were collected at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose from day 1 to day 7, 24 hours post-dose from day 7, day 8 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose. Tmax is a mathematically-derived value from all measurements. Tmax is a measure of the area under the curve that is obtained from plotting the plasma concentration by time point. All time-points were used to derive the single PK parameters.
Time Frame: From pre-dose on day 1 until 12 hours post dose on day 8
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Period 1:Sildenafil;Period 2:LCZ696;Period 3:LCZ696+Sildenafil
Number analyzed (Participants) | 27
hours
  AHU377 | 1.00 (NA) [0.500 to 4.00]
  LBQ657 | 3.00 [1.50 to 6.00]
  valsartan | 2.00 [1.50 to 4.00]

5. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf) of Sildenafil and N-desmethyl-sildenafil Analytes
Description: The effect of co-administration of LCZ696 on the pharmacokinetics of Sildenafil and N-desmethyl-sildenafil was assessed. Blood samples were collected at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose from day 1 to day 7, 24 hours post-dose from day 7, day 8 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose. AUC is a mathematically-derived value from all measurements. AUC is a measure of the area under the curve that is obtained from plotting the plasma concentration by time point. All time-points were used to derive the single PK parameters.
Time Frame: From pre-dose on day 1 until 12 hours post dose on day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Period 1:Sildenafil;Period 2:LCZ696;Period 3:LCZ696+Sildenafil
Number analyzed (Participants) | 27
h*ng/mL
  Sildenafil | 629 (303)
  N-desmethyl-sildenafil | 325 (143)

6. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Sildenafil and N-desmethyl-sildenafil Analytes
Description: as for outcome 5
Time Frame: From pre-dose on day 1 until 12 hours post dose on day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Period 1:Sildenafil;Period 2:LCZ696;Period 3:LCZ696+Sildenafil
Number analyzed (Participants) | 27
h*ng/mL
  Sildenafil | 612 (297)
  N-desmethyl-sildenafil | 305 (133)

7. Primary Outcome: Terminal Elimination Half-life (T1/2) of Sildenafil and N-desmethyl-sildenafil Analytes
Description: The effect of co-administration of LCZ696 on the pharmacokinetics of Sildenafil and N-desmethyl-sildenafil was assessed. Blood samples were collected at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose from day 1 to day 7, 24 hours post-dose from day 7, day 8 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose. T1/2 is a mathematically-derived value from all measurements. T1/2 is a measure of the area under the curve that is obtained from plotting the plasma concentration by time point. All time-points were used to derive the single PK parameters.
Time Frame: From pre-dose on day 1 until 12 hours post dose on day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Period 1:Sildenafil;Period 2:LCZ696;Period 3:LCZ696+Sildenafil
Number analyzed (Participants) | 27
hours
  Sildenafil | 3.84 (1.11)
  N-desmethyl-sildenafil | 6.20 (1.90)

8. Primary Outcome: Maximum Plasma Concentration Following Drug Administration (Cmax) of Sildenafil and N-desmethyl-sildenafil Analytes
Description: The effect of co-administration of LCZ696 on the pharmacokinetics of Sildenafil and N-desmethyl-sildenafil was assessed. Blood samples were collected at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose from day 1 to day 7, 24 hours post-dose from day 7, day 8 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose. All time-points were used to mathematically derive the single PK parameter.
Time Frame: From pre-dose on day 1 until 12 hours post dose on day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Period 1:Sildenafil;Period 2:LCZ696;Period 3:LCZ696+Sildenafil
Number analyzed (Participants) | 27
ng/mL
  Sildenafil | 189 (99.6)
  N-desmethyl-sildenafil | 84.6 (39.3)

9. Primary Outcome: Time to Reach the Maximum Concentration After Drug Administration (Tmax) of Sildenafil and N-desmethyl-sildenafil Analytes
Description: The effect of co-administration of LCZ696 on the pharmacokinetics of Sildenafil and N-desmethyl-sildenafil will be assessed. 8pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose from day 1 to day 7, 24 hours post-dose from day 7, day 8 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose. All time-points were used to mathematically derive the single PK parameter.
Time Frame: From pre-dose on day 1 until 12 hours post dose on day 8
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Period 1:Sildenafil;Period 2:LCZ696;Period 3:LCZ696+Sildenafil
Number analyzed (Participants) | 27
hours
  Sildenafil | 1.00 (NA) [0.500 to 3.00]
  N-desmethyl-sildenafil | 1.00 (NA) [0.500 to 3.00]

10. Secondary Outcome: Adverse Events, Serious Adverse Events and Deaths Were Monitored From Screening to End of Study
Description: Number of patients with adverse events, serious adverse events and death
Time Frame: From the screening visit until 30 days past the final study assessment
Population: Safety Analysis Set: This set included participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Period 1:Sildenafil;Period 2:LCZ696;Period 3:LCZ696+Sildenafil
Number analyzed (Participants) | 28
Participants
  Adverse Events (Serious and non-serious) | 17
  Serious Adverse Events | 0
  Deaths | 0

ADVERSE EVENTS:
Groups:
- Period 1: Sildenafil: During Treatment Period 1, on study Day 1, participants received a single dose of sildenafil followed by wash out on Day 2.
- Period 2: LCZ696: In Period 2 (study Days 3-7), participants received LCZ696 once daily.
- Period 3: LCZ696 + Sildenafil: In Period 3, on study Day 8, participants received LCZ696 , co-administered at the same time with a single dose of sildenafil.
Arm/Group | Period 1: Sildenafil | Period 2: LCZ696 | Period 3: LCZ696 + Sildenafil
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 7/28 | 5/27 | 6/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: Sildenafil (N=28) | Period 2: LCZ696 (N=27) | Period 3: LCZ696 + Sildenafil (N=27)
EYE IRRITATION (Eye disorders) | 2 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 3 | 1
DIZZINESS (Nervous system disorders) | 0 | 2 | 3
HEADACHE (Nervous system disorders) | 3 | 0 | 2
POLLAKIURIA (Renal and urinary disorders) | 0 | 2 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.